CLINICAL TRIAL: NCT05531968
Title: Multicenter, Double-blind, Randomized, Parallel Design, Active-controlled Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of 100 Units of BMI 2006 and Botox® in Adult Patients in Need of Moderate or Severe Glabellar Lines
Brief Title: Treatment of Moderate to Severe Glabellar Lines (BMI2006)
Acronym: BMI2006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BMI Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMI2006-SIT-02
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Glabellar Lines
Keywords: BMI2006; BMI; Botulinum toxin; Clostridium botulinum Type A; BOTOX; BoNT-A; corrugator supercilii muscle
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI2006 100Units (Experimental): Patients were intramuscularly injected (IM) with a total of 20U of BMI2006 in 5 places of 0.1 mL (4 U/0.1 mL) each on the glabellar line.
  Interventions: Biological: BMI2006
- Botox® (Active Comparator): Patients were intramuscularly injected (IM) with a total of 20U of Botox® in 5 places of 0.1 mL (4 U/0.1 mL) each on the glabellar line.
  Interventions: Biological: BOTOX®

INTERVENTIONS:
Biological: BMI2006 — IM
  Other Names: Clostridium botulinum Type A
  Arms: BMI2006 100Units
Biological: BOTOX® — IM
  Other Names: Clostridium botulinum Type A
  Arms: Botox®

SUMMARY:
A multicenter, double-blind, randomized, parallel design, active control, phase 3 clinical trial to evaluate the efficacy and safety of 100 units of BMI 2006 and Botox® in adult patients in need of moderate or severe glabellar lines

DETAILED DESCRIPTION:
Purpose of clinical trial:

The purpose of this study was to evaluate the efficacy and safety of 20U dose administration of 100 units of BMI2006 in adult patients who needed moderate or severe glabellar lines.

primary purpose Comparing the effectiveness after administration of each 20U dose of 'BMI2006 100 Units' or 'Botox® Week' for adult patients in need of moderate or severe glabellar lines, it was found that the BMI2006 injection group was non-inferior to the Botox® injection group. wanted to confirm.

secondary purpose The purpose of this study was to evaluate the safety and effectiveness of 'BMI2006 100 Units' 20U compared to 'Botox® Injection' 20U for adult patients who need moderate or severe glabellar wrinkles.

This clinical trial was designed as a multicenter, double-blind, randomized, parallel design, active-controlled Phase 3 clinical trial, and was intended for patients with moderate or severe glabellar lines.

Only those subjects who have agreed in writing to voluntarily participate in the clinical trial and who are evaluated to meet the selection/exclusion criteria are 1:1 to the test group (BMI2006 week administration group) or control group (Botox®) in the order of participation in the clinical trial was randomly assigned.

Subjects assigned with randomization numbers were intramuscularly injected (IM) with a total of 20U of clinical trial drugs in 5 places of 0.1 mL (4 U/0.1 mL) each on the glabellar line. Thereafter, at 4, 8, 12, and 16 weeks at intervals of 4 weeks, the institution was visited to evaluate the efficacy and safety for a total of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged between 19 and 65
2. Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
3. Patients who fully understand the clinical trial and voluntarily sign the informed consent

Exclusion Criteria:

1. Patients with neuromuscular junction disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis[ALS], etc.)
2. Patients with facial palsy or blepharoptosis
3. Patients who have marked facial asymmetry
4. Patients whose glabellar lines cannot be satisfactorily improved with physical method since the lines are not flattened even using hands
5. Patients who have received the medications that cause relaxation of muscles all over the body within 4 weeks prior to screening

   * Muscle Relaxants (e.g., Tubocurarine chloride, Dantrolene sodium, Baclofen, etc.)
   * Spectinomycin hydrochloride
   * Aminoglycoside antibiotics (e.g., Gentamicin sulfate, Neomycin sulfate, etc.)
   * Polypeptide antibiotics (e.g., Polymyxin B sulfate, etc.)
   * Tetracycline antibiotics
   * Lincosamide antibiotics
   * Aanticholinergic agent (e.g., Butylscopolamine bromide, Trihexyphenidyl hydrochloride, etc.)
   * Benzodiazepines (e.g., Diazepam, Etizolam, etc.)
   * Other medications that cause relaxation of muscles all over the body
6. Patients who have received anticoagulant, antiplatelet agent or NSAIDs within 7 days before the first dose (Allow use of low-dose Aspirin[325 mg/day or less] for the antithrombotic therapy)
7. Patients with skin disorders, infection or scars at the injection site
8. Patients who have received other procedures which may affect glabellar and forehead lines within 12 months prior to screening

   * Permanent soft tissue augmentation (e.g., Permanent filler, etc.)
   * Face lifting (e.g., Forehead/Browlift, Thread lifting, etc.)
   * Implant and Fat grafting
9. Patients with the history of treatment of glabellar part(including forehead) which may affect the treatment results

   * Hyaluronic Acid/Collagen fillers, Dermal resurfacing, Chemical Peeling, dermabrasion and Dermal Photorejuvenation within 6 months
   * Dermer Filler and Nonpermanent soft tissue filler within 12 months
10. Patients who have a plan to receive facial cosmetic procedures including dermal filler, photorejuvenation, chemical peeling and dermabrasion during the study period
11. Patients who have a history of injecting drugs similar to the investigational drugs within 6 months prior to selection or are foreseen to use Botulinum Toxin A type or Botulinum Toxin B type during the study period
12. Patients who have received Retinoids (e.g., isotretinoin, alitretinoin, etc.)

    * Systemic agents: within 6 months prior to screening
    * Topical agents: within 3 months prior to screening
13. Patients with the history of alcohol or drug addiction
14. Patients who have anxiety or mental disorder (e.g., depression) which may affect patient participation or objective efficacy assessment results based on the judgment of an investigator
15. Fertile women and men who have a plan on being pregnant during the study or are not willing to use appropriate contraception
16. Pregnant or lactating women
17. Patients with allergy or hypersensitivity to the investigational drugs or their components
18. Patients who have a disorder associated with malignant tumor, immunodeficiency(weak immune system), kidney disease, liver disease lung disease or etc., which is unsuitable for participation of the study based on the judgment of an investigator
19. Patients who have participated in other clinical trials and were received or applied with other investigational products or investigational device within 30 days prior to screening
20. Patients whom the investigator judges to be unsuitable to participate

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Change rate of glabellar line at maximum frown confirmed with investigator's on-site assessment of FWS | 0 and 4 weeks after the injection
  Change rate of glabellar line at maximum frown confirmed with investigator's on-site assessment of Facial Wrinkle Scale at baseline and 4 weeks after the injection

SECONDARY OUTCOMES:
Change rate of glabellar line at maximum frown confirmed with investigator's on-site assessment of FWS | 0, 8, 12 and 16 weeks after the injection
  Change rate of glabellar line at maximum frown confirmed with investigator's on-site assessment of Facial Wrinkle Scale at baseline, 8, 12 and 16 weeks after the injection
Change rate of glabellar line at rest confirmed with investigator's on-site assessment of FWS | 0, 4, 8, 12 and 16 weeks after the injection
  Change rate of glabellar line at rest confirmed with investigator's on-site assessment of Facial Wrinkle Scale at baseline, 4, 8, 12 and 16 weeks after the injection
Change rate of glabellar line at maximum frown confirmed with independent evaluator's photo assessment of FWS | 0, 4, 8,12 and 16 weeks after the injection
  Change rate of glabellar line at maximum frown confirmed with independent evaluator's photo assessment of Facial Wrinkle Scale at baseline, 4, 8,12, 16 weeks after the injection
Change rate of glabellar line at rest confirmed with independent evaluator's photo assessment of FWS | 0, 4, 8,12 and 16 weeks after the injection
  Change rate of glabellar line at rest confirmed with independent evaluator's photo assessment of Facial Wrinkle Scale at baseline, 4, 8,12, 16 weeks after the injection
Change rate of glabellar line confirmed with subject's assessment of the Subject Questionnaire | 4, 8, 12 and 16 weeks after the injection
  Change rate of glabellar line confirmed with subject's assessment of the Subject Questionnaire that underpin the nine-scale change of glabellar line at 4, 8, 12 and 16 weeks after the injection
Satisfaction level using the Subject Satisfaction Questionnaire | 4, 8, 12 and 16 weeks after the injection
  Satisfaction level using the Subject Satisfaction Questionnaire that underpin the seven-scale measurement of satisfaction at 4, 8, 12 and 16 weeks after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, MD, Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (3):
- South Korea (3):
  - Chung-Ang University Hospital, Seoul, Heukseok-ro, Dongjak-gu
  - Konkuk University Hospital, Seoul, Neungdong-ro, Gwangjin-gu
  - Seoul Asan Medical Center, Seoul, Olympic-ro 43-gil, Songpa-gu